CLINICAL TRIAL: NCT00521456
Title: A Study of Ketorolac for the Treatment of Inflammation and Pain Associated With Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 191578-006
Record Dates: First submitted 2007-08-23; First posted 2007-08-27 (Estimated); Results first posted 2009-10-01 (Estimated); Last update posted 2009-10-01 (Estimated); Status verified 2009-08

CONDITIONS: Cataract Extraction

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: ketorolac eye drops
- 2 (Placebo Comparator)
  Interventions: Drug: ketorolac eye drops

INTERVENTIONS:
Drug: ketorolac eye drops — 1 drop twice daily day preop and Days 1-14, and 6 doses on surgery day
  Placebo

SUMMARY:
This is a 16 day study to evaluate the safety and efficacy of ketorolac eye drops for the treatment of inflammation and pain associated with cataract surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cataract surgery

Exclusion Criteria:

* Uncontrolled ocular disease in cataract surgery eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2007-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- San Diego, California, United States

REFERENCES:
- [Derived] Donnenfeld ED, Nichamin LD, Hardten DR, Raizman MB, Trattler W, Rajpal RK, Alpern LM, Felix C, Bradford RR, Villanueva L, Hollander DA, Schiffman RM. Twice-daily, preservative-free ketorolac 0.45% for treatment of inflammation and pain after cataract surgery. Am J Ophthalmol. 2011 Mar;151(3):420-6.e1. doi: 10.1016/j.ajo.2010.09.003. Epub 2010 Dec 9. PMID 21145532
- See also: Related Info — http://www.allerganclinicaltrials.com/inquiries/trialsubject.aspx

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketorolac Solution | Vehicle Solution
Started | 176 | 87
Completed | 163 | 59
Not Completed | 13 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketorolac Solution | Vehicle Solution | Total
Number analyzed (Participants) | 176 | 87 | 263
Age, Customized [Number; unit: participants]
  <45 years | 4 | 3 | 7
  Between 45 and 65 years | 56 | 32 | 88
  >65 years | 116 | 52 | 168
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 51 | 152
  Male | 75 | 36 | 111

OUTCOME MEASURES:

1. Primary Outcome: Resolution of Post Operative Inflammation
Description: Anterior chamber inflammation is the sum of biomicroscopic cell and flare; each measured on a scale of 0-4 (Flare: 0 = no flare, 4 = intense flare / Cell: 0 = no cells, 4 = >50 cells)
Time Frame: Day 14
Population: Modified Intent-to-Treat Population
Measure: Number; unit: % of participants with a score of 0
Arm/Group | Ketorolac Solution | Vehicle Solution
Number analyzed (Participants) | 169 | 77
% of participants with a score of 0 | 58.0 | 27.3

2. Secondary Outcome: Ocular Pain
Description: Measured on a scale of 0-4 (0 = none, 4 = intolerable)
Time Frame: Day 1
Population: Modified Intent-to-Treat Population
Measure: Number; unit: % of participants with a score of 0
Arm/Group | Ketorolac Solution | Vehicle Solution
Number analyzed (Participants) | 170 | 78
% of participants with a score of 0 | 70.0 | 38.5

3. Secondary Outcome: Mean Pupil Area
Description: Pupil area post-irrigation and aspiration
Time Frame: Day 0
Population: Modified Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: millimeters squared (mm²)
Arm/Group | Ketorolac Solution | Vehicle Solution
Number analyzed (Participants) | 173 | 81
millimeters squared (mm²) | 37.9 (12.0) | 36.5 (13.5)

4. Post Hoc Outcome: Visual Acuity
Description: Patients with ≥ 3 line improvement in visual acuity
Time Frame: Change from baseline at Day 14
Population: Modified Intent-to-Treat Population
Measure: Number; unit: Percentage of patients with ≥ 3 lines
Arm/Group | Ketorolac Solution | Vehicle Solution
Number analyzed (Participants) | 167 | 80
Percentage of patients with ≥ 3 lines | 56.9 | 36.3

ADVERSE EVENTS:
Arm/Group | Ketorolac Solution | Vehicle Solution
Serious Adverse Events (participants affected / at risk) | 1 | 0
Other Adverse Events (participants affected / at risk) | 68 | 57
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Ketorolac Solution | Vehicle Solution
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1/173 | 0/82
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Ketorolac Solution | Vehicle Solution
Conjunctival Hyperaemia (Eye disorders) | 12/173 | 11/82
Anterior chamber cell (Eye disorders) | 12/173 | 6/82
Anterior chamber flare (Eye disorders) | 11/173 | 6/82
Corneal edema (Eye disorders) | 9/173 | 8/82
Eye pain (Eye disorders) | 7/173 | 10/82
Iritis (Eye disorders) | 6/173 | 7/82
Photophobia (Eye disorders) | 1/173 | 8/82
Intraocular pressure increased (Investigations) | 10/173 | 1/82

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.